CLINICAL TRIAL: NCT04249115
Title: Prospective, Open-Label, Multi-Center, Non-Significant Risk Study of Nano-Pulse Stimulation™ (NPS™) Technology in Healthy Adults With Seborrheic Keratosis
Brief Title: Nano-Pulse Stimulation (NPS) in Seborrheic Keratosis Optimization Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment was halted due to a business decision by the Sponsor to focus resources on other clinical areas outside of dermatology.
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-SK-008
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Lesion Skin; Seborrheic Keratosis; Skin Lesion; Benign Skin Tumor
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Nano-Pulse Stimulation (NPS) Treated Lesion (Experimental): Nano-Pulse Stimulation of targeted lesion.
  Interventions: Device: Nano-Pulse Stimulation (NPS)

INTERVENTIONS:
Device: Nano-Pulse Stimulation (NPS) — Electrical pulses (nanosecond duration) applied directly to target SK lesions using sterile single-patient use treatment tips with microneedles.

SUMMARY:
Primary study objective is to evaluate the optimization of Nano-Pulse Stimulation (NPS) energy settings for lesion clearance of Seborrheic Keratosis (SKs) from off-facial areas of healthy adults.

DETAILED DESCRIPTION:
* Evaluate lesion clearance rate of SKs in off-face locations post-treatment versus baseline using multiple sized treatment tips with microneedles.
* Evaluate the clearance of the treated SKs using multiple energy settings at various time points initial procedure, compared baseline.
* Evaluate skin effects and adverse event rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 21 and 75 years of age
* Voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained
* Understanding of the clinical investigation, agree to cooperate with the investigational procedures and willing to return for all the required follow-up visits
* Understands that SKs are to be treated in a single treatment session and is aware that they may receive a second treatment
* Must be able to visit clinic site at 7-, 30-, 60-, and 90-days post-primary treatment of SK lesion and at retreatment
* Clinical diagnosis of stable, clinically typical Seborrheic Keratosis
* Minimum of two SK lesions
* SKs must be no greater than 2mm in height and not exceed 10mm x 10mm at their largest point
* Undergo all study procedures including consent for global photographs of the SK study sites
* Agrees to refrain from using all other SK lesion removal products or treatments (topical medication including over-the-counter medications) during the study period

Exclusion Criteria:

* Implantable electronic devices (i.e., automatic defibrillator)
* Active infection or history of infection in designated test area within 90 days prior to first treatment
* Not willing or able to sign the Informed Consent
* Known to be immune-compromised
* Known to be keloid producer
* Taking blood thinning medications
* Insulin dependent, Type I diabetics
* Allergies to Lidocaine or Lidocaine-like products
* Employed by the sponsor, clinic site, or entity associated with the conduct of the study
* Family member of someone employed by the sponsor, clinic site, or entity associated with the conduct of the study
* Have any condition or situation which, in the Investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study
* Prior inability to complete required study visits during treatment period.
* Use of any other investigational drug, therapy, or device within the past 30 days of enrollment or concurrent participation in another research study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Clearance Rate of SK Lesions | 90 days post-last treatment
  Degree of Clearance of SK lesion treated with NPS as rated by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (7):
- United States (7):
  - Clear Dermatology & Aesthetics Center / InvestigateMD, Scottsdale, Arizona
  - Mountain Dermatology Specialists, Edwards, Colorado
  - SKIN Associates of South Florida, Coral Gables, Florida
  - Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - Zel Skin & Laser Specialists, Edina, Minnesota
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No